CLINICAL TRIAL: NCT01827059
Title: A Randomized Placebo Controlled Trial to Analyze Changes in Pulmonary Arterial Pressures at Peak Exercise in Congenital Heart Disease Patients With Exercise-induced Pulmonary Arterial Hypertension Before and After Treatment With Bosentan, Compared to Placebo
Brief Title: Bosentan In Exercise Induced Pulmonary Arterial Hypertension in CongenitaL Heart diseasE
Acronym: BICYCLE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Berto J Bouma, Dr. B.J. Bouma, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL 42568.018.12
Record Dates: First submitted 2013-04-05; First posted 2013-04-09 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Arterial Hypertension; Congenital Heart Disease
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Heart Defects, Congenital | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bosentan (Active Comparator): Tracleer, 125-mg orange-white, round, biconvex, film-coated tablets
  Interventions: Drug: Bosentan
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bosentan — 125-mg orange-white, round, biconvex, film-coated tablets
  Other Names: Tracleer
  Arms: Bosentan
Drug: Placebo
  Arms: Placebo

SUMMARY:
SUMMARY Rationale: Pulmonary arterial hypertension (PAH) can be a rapidly progressive disorder and is associated with a high mortality rate, despite medical intervention. With the availability of effective therapy, early disease detection is an important strategic objective to improve treatment outcomes. Resting echocardiography is currently the recommended screening modality for high-risk population groups. However, it is clear that abnormalities in resting hemodynamics (and symptoms) are late sequelae of the pathobiological processes that begin in the distal pulmonary arteries. Exercise stress may unmask early pulmonary vascular dysfunction, however the definition, clinical significance, and natural history of 'exercise PAH' remain undefined. However, based on clinical experience and literature the prevalence is estimated at ~ 20%.Treatment with endothelin receptor blockers has shown a beneficial influence on the clinical performance in patients with exercise induced PAH due to systemic sclerosis and primary pulmonary hypertension. Whether endothelin receptor blockers decrease pulmonary pressures and improve clinical outcome in patients with exercise induced pulmonary arterial hypertension due to congenital heart disease is unknown.

Objective: Identify congenital heart disease patients with exercise-induced pulmonary arterial hypertension. Analyze changes in pulmonary arterial pressures at peak exercise in patients with exercise induced pulmonary arterial hypertension before and after treatment with bosentan, compared to placebo.

Study design: Randomized placebo controlled trial with a study period of 26 weeks.

Study population: Adult congenital heart disease patients with exercise induced pulmonary arterial hypertension (n=40) from the Academic Medical Centre, Amsterdam.

Intervention: After randomization one group (n=20) receives a 125 mg tablet of Bosentan twice daily for 6 months. The other group (n=20) receives placebo for 6 months.

Main study parameters/endpoints: To determine wether bosentan (endothelin receptor inhibitor) decreases mean pulmonary arterial pressure at peak exercise in adult congenital heart disease patients with exercise induced pulmonary arterial hypertension. Furthermore the change in cardiopulmonary exercise capacity and right ventricular function will be investigated.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All investigations, blood analysis excepted, are non-invasive and free of risk. The burden for the patients mainly consists of the time that is consumed by the investigations, namely: history taking + physical examination (15 min); Quality-of-Life- score (15 min); laboratory tests (electrolytes, creatinine, urea, albumin and neurohormones, troponin T); 12 lead electrocardiogram (10 min); exercise echocardiography (30 min); cardiovascular exercise testing (30 min).

The trial medication has a potential risk of liver damage, which will be monitored regularly by laboratory testing of liver transaminases.

ELIGIBILITY:
Inclusion Criteria:

* adult (>18 years) and mentally competent
* Open or closed septal defect (ASD I/II, VSD, AVSD)
* Open or closed systemic-to-pulmonary shunt (PDA, PAPVC)
* Negative pregnancy test
* Presence of X-PAH

  * One of the following criteria, at peak exercise.
  * mPAP > 34 mmHg with CO ≤ 10 l/min
  * mPAP > 40 mmHg with CO ≤ 15 l/min
  * mPAP > 45 mmHg with CO ≤ 20 l/min
  * mPAP > 50 mmHg with CO ≤ 30 l/min
  * a PVR (slope pressure/flow plot) of > 3 mmHg/l/min

Exclusion Criteria:

* Incapable of giving informed consent
* Pregnancy or lactation (a pregnancy test is offered to every female patient within fertile age)
* Women of child-bearing age who are sexually active without practising reliable methods of contraception. The use of oral contraceptives only, is not considered reliable. Reliable methods include concomitant use of oral contraceptives and condoms ("Double Dutch"), and those methods with a less than 1% chance of pregnancy during typical use20, including intrauterine contraceptives (Copper T, Mirena), Implanon, and sterilization.
* Substance abuse (alcohol, medicines, drugs)
* Subjects who are not able to perform cardiopulmonary exercise testing
* Any cardiac operation < 6 months before inclusion
* PAH of any aetiology other than the one specified in the inclusion criteria
* Left ventricular ejection fraction < 30%
* Significant impairment of renal function (GFR < 30 ml/min/1.73m2)
* Moderate to severe liver disease: Child Pugh class B or C
* Raised plasma transaminases level > three times upper normal limit
* Arterial hypotension (systolic blood pressure < 85mmHg)
* Anaemia (Hb < 10g/L, or <6.21 mmol/L)
* Significant valvular disease, other than tricuspid or pulmonary regurgitation
* Chronic lung disease or total lung capacity < 80% predicted value
* History of significant pulmonary embolism
* Other relevant diseases (HIV infection, Hep B/C infection)
* Subjects with known intolerance to bosentan or their constituents
* Prohibited medication: any medication listed below which has not been discontinued at least 30 days prior to inclusion

  * Unspecified or other significant medication (glibenclamide or immunosuppression)
  * PAH therapy (endothelin receptor antagonists, PDE-5 inhibitors, prostanoids)
  * Medication which is not compatible with bosentan or interferes with its metabolism (inhibitors or inducers of CYP2C9, CYP3A4) or medication which may interfere with bosentan treatment according to the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-10; Primary Completion 2018-02 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change in mean pulmonary arterial pressure (mPAP) at peak exercise | 26 weeks
  * measured by means of transthoracic echocardiography at 3 and 6 months followup: mPAP = 0.6 x systolic PAP.
  * peak exercise is defined as 80% of maximum calculated heart rate: peak exercise=0.8*(220-age)

SECONDARY OUTCOMES:
Cardiopulmonary exercise capacity | 26 weeks
  o i.e. peak oxygen consumption, VE/VCO2 ratio, O2 pulse
Pulmonary hemodynamics | 26 weeks
  o i.e. systolic pulmonary arterial pressure, pulmonary vascular resistance, pressure-flow relationships during and at peak exercise
Right ventricular function | 26 weeks
  o i.e. TAPSE, TEI index, TDI-S, right ventricular dimensions
Laboratory parameters | 26 weeks
  o i.e. NT-pro BNP, troponin T
NYHA functional class | 26 weeks
Quality of life | 26 weeks
  o assessed by TAAQOL-CHD, SF-36 and Minnesota CHD-HF questionnaire
Demographics | 26 weeks
  * age, gender, marital status, work, income.
  * assessed by demographic questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: A.C.J.M. van Riel, MD, Principal Investigator — Academic Medical Centre; B.J. Bouma, MD, PhD, Principal Investigator — Academic Medical Centre; B.J.M. Mulder, MD, PhD, Principal Investigator — Academic Medical Centre
Locations (1):
- Academic Medical Centre, Amsterdam, North Holland, Netherlands